CLINICAL TRIAL: NCT05371314
Title: Artificial Intelligence in Categorizing the Severity of Oxygenation by Incorporating the PEEP Into the Definition of ARDS in Ventilated Patients
Acronym: P/FP ratio
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Sunitha PalaniDurai, Principal Investigator, National University Health System, Singapore
Other Study IDs: NUHS
Record Dates: First submitted 2022-05-02; First posted 2022-05-12 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: ARDS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: P/FP ratio — PaO2/FiO2 X PEEP, SpO2/FiO2 X PEEP

SUMMARY:
Artificial Intelligence in categorizing the severity of Oxygen in ventilated patients to predict initiation of treatment measures to improve mortality - P/FP ratio

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients

Exclusion Criteria:

1. pediatric and neonates
2. DNR patients
3. Non intubated patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from MIMIC 4 and eICU
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Artificial intelligence in categorizing the severity of oxygenation of ARDS in ventilated patients | Baseline ABG done at (approximately 4 hour after intubation) to ABG done day 2,3 and day 7
  To see the trend and difference between day 1, 2,3 and day 7 between P/F (PaO2/FiO2) and S/F(SaO2/FiO2) ratio to P/FP (PaO2/FiO2*PEEP) ratio and S/FP (SpO2/(FiO2*PEEP) ratio respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- National Universty Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No